CLINICAL TRIAL: NCT02065895
Title: Effect of Gain on Closed-Loop Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P-000401
Record Dates: First submitted 2014-02-07; First posted 2014-02-19 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes
Keywords: Physiologic Insulin Delivery (PID); Closed Loop; Sensor; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Medication Errors

STUDY DESIGN:
Intervention Model Description: Study subjects are studied under closed-loop control on three occasions: once with the glucose values used for control equal to blood glucose (NO error), once with values 33% higher than blood glucose (HIGH error), and once with values 20% lower than blood glucose (LOW error). The six different sequences of these three exposures then comprise the six arms of this crossover study.
Oversight: Data Monitoring Committee: No

ARMS (6):
- HIGH error, LOW error, NO error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with glucose-value-used-for-control higher than blood glucose (HIGH error), then second with glucose-value-used-for-control lower than blood glucose (LOW error), then third with glucose-value-used-for-control equal blood glucose (NO error).
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error
- HIGH error, NO error, LOW error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with glucose-value-used-for-control higher than blood glucose (HIGH error), then second with glucose-value-used-for-control equal blood glucose (NO error), then third with glucose-value-used-for-control lower than blood glucose (LOW error).
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error
- NO error, HIGH error, LOW error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with glucose-value-used-for-control equal blood glucose (NO error), then second with glucose-values-used-for-control higher than blood glucose (HIGH error), then third with glucose-value-used-for-control lower than blood glucose (LOW error).
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error
- NO error, LOW error, HIGH error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with glucose-value-used-for-control equal blood glucose (NO error), then second with glucose-value-used-for-control lower than blood glucose (LOW error), then third with glucose-value-used-for-control higher than blood glucose (HIGH error).
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error
- LOW error, NO error, HIGH error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with with glucose-value-used-for-control lower than blood glucose (LOW error), then second with glucose-value-used-for-control equal blood glucose (NO error), then third with glucose-value-used-for-control higher than blood glucose (HIGH error).
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error
- LOW error, HIGH error, NO error (Experimental): Subjects were randomized to receive overnight and breakfast closed-loop glucose control glucose on three occasions: first with glucose-value-used-for-control lower than blood glucose (LOW error), then second with glucose-value-used-for-control equal blood glucose (NO error), then third glucose-value-used-for-control higher than blood glucose (HIGH error),
  Interventions: Device: HIGH error; Device: NO error; Device: LOW error

INTERVENTIONS:
Device: HIGH error — Overnight and breakfast closed-loop control were performed using a target glucose of 120 mg/dL but with the glucose-value-used-for-control equal to 1.33 times the true glucose value (analogous to higher gain lower target).
Device: NO error — Overnight and breakfast closed-loop control were performed using a target glucose of 120 mg/dL and glucose-value-used-for-control equal to the true glucose value.
Device: LOW error — Overnight and breakfast closed-loop control were performed using a target glucose of 120 mg/dL but with the glucose-value-used-for-control equal to 0.8 times the true glucose value (analogous to lower gain higher target).

SUMMARY:
The purpose of this study is to test the ability of an advanced external Physiologic Insulin Delivery (ePID) algorithm (a step by step process used to develop a solution to a problem) to get acceptable meal responses over a range of gain. Gain is defined as how much insulin is given in response to a change in a patient's glucose level.

This study also examines the effectiveness of the external Physiologic Insulin Delivery (ePID) closed-loop insulin delivery computer software. The investigators would like to assess whether fasting target levels can be achieved as the closed-loop gain increases or decreases, and to evaluate the system's ability to produce an acceptable breakfast meal response.

DETAILED DESCRIPTION:
There have been significant advances in diabetes management technology, including more sophisticated insulin pumps and more accurate real-time continuous glucose monitors. The next technological development is widely thought to be the introduction of an algorithm linking the pump and sensor to form a closed-loop insulin delivery system. The algorithm used for this purpose needs to be robust to changes in an individual's insulin sensitivity, and the sensor's sensitivity to glucose. Insulin sensitivity (how much the patient's glucose level changes in response to a change in insulin delivery) and algorithm gain (how much insulin is delivered in response to a change in glucose) determine the systems overall closed-loop gain. Ideally, the overall gain can be set to achieve the lowest possible peak postprandial glucose response without postprandial hypoglycemia. However, if the algorithm's gain is set to a fixed value and the subject's insulin sensitivity changes, the overall-gain will change. Some degradation in closed-loop performance might be acceptable during periods whenever the subject's insulin sensitivity is low (i.e., the subject is insulin resistant) and the risk of hypoglycemia may actually be reduced. However, if the subject becomes more sensitive the system may become less stable and the risk of postprandial hypoglycemia may increase. In addition to changes in insulin sensitivity, glucose sensors will sometimes over- or under-read blood glucose as sensor sensitivity increases or decreases. This will result in a change in the closed-loop algorithm's effective target. The purpose of this study is to evaluate the ability of an advanced Physiologic Insulin Delivery algorithm to achieve an acceptable breakfast response as the gain and effective target glucose level changes. Specifically:

1. to assess the fasting glucose levels achieved as the overall closed-loop gain and effective target is increased or decreased, and
2. determine the system's ability to produce an acceptable breakfast meal response under these conditions

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for > 3 years
* Manage diabetes using a continuous glucose monitor and continuous subcutaneous insulin infusion pump
* Non obese (BMI < 30)
* Aged 18 - 75 years old
* HbA1c < 8 %

Exclusion Criteria:

* renal or hepatic failure
* cancer or lymphoma
* Malabsorption or malnourishment
* Hypercortisolism
* Alcoholism or drug abuse
* Anemia (hematocrit < 36 in females and <40 in males)
* Eating disorder
* Dietary restrictions
* Acetaminophen allergy
* Chronic acetaminophen use
* Glucocorticoid therapy
* History of gastroparesis
* Use of Beta blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steil GM, Panteleon AE, Rebrin K. Closed-loop insulin delivery-the path to physiological glucose control. Adv Drug Deliv Rev. 2004 Feb 10;56(2):125-44. doi: 10.1016/j.addr.2003.08.011. PMID 14741112
- [Background] Steil GM, Rebrin K, Janowski R, Darwin C, Saad MF. Modeling beta-cell insulin secretion--implications for closed-loop glucose homeostasis. Diabetes Technol Ther. 2003;5(6):953-64. doi: 10.1089/152091503322640999. PMID 14709197
- [Background] Steil GM, Rebrin K, Darwin C, Hariri F, Saad MF. Feasibility of automating insulin delivery for the treatment of type 1 diabetes. Diabetes. 2006 Dec;55(12):3344-50. doi: 10.2337/db06-0419. PMID 17130478
- [Background] Weinzimer SA, Steil GM, Swan KL, Dziura J, Kurtz N, Tamborlane WV. Fully automated closed-loop insulin delivery versus semiautomated hybrid control in pediatric patients with type 1 diabetes using an artificial pancreas. Diabetes Care. 2008 May;31(5):934-9. doi: 10.2337/dc07-1967. Epub 2008 Feb 5. PMID 18252903
- [Background] Steil GM, Palerm CC, Kurtz N, Voskanyan G, Roy A, Paz S, Kandeel FR. The effect of insulin feedback on closed loop glucose control. J Clin Endocrinol Metab. 2011 May;96(5):1402-8. doi: 10.1210/jc.2010-2578. Epub 2011 Mar 2. PMID 21367930
- [Background] Loutseiko M, Voskanyan G, Keenan DB, Steil GM. Closed-loop insulin delivery utilizing pole placement to compensate for delays in subcutaneous insulin delivery. J Diabetes Sci Technol. 2011 Nov 1;5(6):1342-51. doi: 10.1177/193229681100500605. PMID 22226251
- [Background] Buchanan TA, Xiang AH, Peters RK, Kjos SL, Berkowitz K, Marroquin A, Goico J, Ochoa C, Azen SP. Response of pancreatic beta-cells to improved insulin sensitivity in women at high risk for type 2 diabetes. Diabetes. 2000 May;49(5):782-8. doi: 10.2337/diabetes.49.5.782. PMID 10905487
- [Background] Panteleon AE, Loutseiko M, Steil GM, Rebrin K. Evaluation of the effect of gain on the meal response of an automated closed-loop insulin delivery system. Diabetes. 2006 Jul;55(7):1995-2000. doi: 10.2337/db05-1346. PMID 16804068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Written informed consent was obtained from all 8 participants at the Joslin Diabetes Center. All study related activities were conducted at the Center for Clinical Investigations at the Beth Israel deaconess Medical Center.
Groups:
- HIGH Error First, LOW Error Second, Then NO Error Third: In this arm, subjects were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control calculated to be 33% higher than the true glucose value (HIGH error), then second with the value calculated to be 20% lower than the true value (LOW error), then third with the value equal to the true value (NO error). These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes). Intervention period: 17 hours; minimum washout period was 7 hours, maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
- HIGH Error First, NO Error Second, Then LOW Error Third: In this arm, subjects were were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control calculated to be 33% higher than the true glucose value (HIGH error), then second with the value calculated to equal the true value (NO error), and then third with the value calculated to be 20% lower than the true value (LOW error). These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes). Intervention period: 17 hours; minimum washout period was 7 hours, maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
- NO Error First, LOW Error Second, HIGH Error Third: In this arm, subjects were were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control equal the true value (NO error), then second with the value calculated to be 20% lower than the true value (LOW error), and then third with the value calculated to be 33% higher than the true glucose value (HIGH error). These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes). Intervention period: 17 hours; minimum washout period was 7 hours, maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
- NO Error First, HIGH Error Second, LOW Error Third: In this arm, subjects were were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control calculated equal the true value (NO error), and then second with the value calculated as 33% higher than the true glucose value (HIGH error), and then third with the value calculated to to be 20% lower than the true glucose value (LOW error). These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes).Intervention period: 17 hours; minimum washout period was 7 hours, maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
- LOW Error First, NO Error Second, HIGH Error Third: In this arm, subjects were were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control calculated to be 20% lower than the true glucose value (LOW error), then second with the value calculated to equal the true value (NO error), and then third with the value calculated to be 33% higher than the true value. These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes). Intervention period: 17 hours; minimum washout period was 7 hours,maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
- LOW Error First, HIGH Error Second, NO Error Third: In this arm, subjects were were randomized to undergo in-clinic closed-loop control of nighttime and breakfast glucose on three occasions: first with the glucose value used for control calculated to be 20% lower than the true glucose value (LOW error), then second with the value calculated to be 33% higher than the true value (HIGH error), and then third with the value calculated to be equal the true value (NO error). These conditions reflect real-life conditions that would be expected if closed-loop artificial pancreas control is effected with different sensor calibration error. No meal announcement was provided (simulates condition where patient forgets to announce meal), and all subjects were controlled with the same closed-loop gain (simulates conditions where an individual's insulin sensitivity changes). Intervention period: 17 hours; minimum washout period was 7 hours, maximum was 62 days (varied among subjects, allowed up to 3 months to complete all 3 interventions).
Period: Overall Study
Arm/Group | HIGH Error First, LOW Error Second, Then NO Error Third | HIGH Error First, NO Error Second, Then LOW Error Third | NO Error First, LOW Error Second, HIGH Error Third | NO Error First, HIGH Error Second, LOW Error Third | LOW Error First, NO Error Second, HIGH Error Third | LOW Error First, HIGH Error Second, NO Error Third
Started | 1 | 3 | 1 | 1 | 1 | 1
Completed | 0 | 2 | 1 | 0 | 1 | 1
Not Completed | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Scheduling conflicts | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject withdrew prior to visit 1; of the seven subjects admitted on 3 occasions, two had protocol violations on one occasion (one subject experienced technical problems; one subject completed the nighttime period but was called away on an emergency prior to breakfast); 5 subjects completed the study per protocol.
Groups:
- Closed-loop Control: Closed-loop control was performed from 9:00 PM to 2:00 the day following admission on three occasions: once with a glucose-value-used-for control calculated to be higher than the true blood glucose (analogous to a sensor glucose signal that is miss-calibrated); once with the value equal to blood glucose (analogous to a sensor signal with no calibration), and once with the value calculated to be lower than blood glucose. Six different arms were utilized, defined by the differing sequences of each of the three values used for control (no error, high error and low error previously defined). On each occasion control was separated into the nighttime period (midnight to 08:00 AM) and breakfast period (8:00 AM to 2:00 PM).
Arm/Group | Closed-loop Control
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 57 [40 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants] — Population: One subject withdrew
  participants
    United States | 8
Median duration of diabetes [Median (Full Range); unit: years] | 47 [11 to 62]
Daily insulin use [Mean (Full Range); unit: units/day] | 35.4 [27 to 45.2]
HbA1c [Mean (Full Range); unit: %] | 7.7 [6.8 to 8.4]

OUTCOME MEASURES:

1. Primary Outcome: Glucose Area Under the Curve (AUC) Breakfast
Description: Glucose Area Under the Curve (AUC) Breakfast defines the total exposure to glucose during breakfast. Breakfast is typically considered the most difficult meal to control; low AUC is desirable.This outcome measure was analyzed for each of the three calibration error values (high error, no error and low error).
Time Frame: On day #1, day #2 and day #3 (each day could be 24 hours to 7 days apart from prior one, and completed within 6 week period) 8:00 AM to 2:00 PM on day following admission, with samples obtained every 10-15 minutes, for each sequence of calibration errors
Measure: Mean (95% Confidence Interval); unit: mmol/l/min
Groups:
- HIGH Error: Glucose sensor errors leading to sensor glucose reading higher than that true blood glucose result in closed-loop control systems (artificial pancreas) behaving as if the control gain is increased and the target is lowered. In this arm we study closed-loop control with a sensor signal reading 33% higher than blood glucose.
- NO Error: Glucose sensor errors leading to sensor glucose reading higher than that true blood glucose result in closed-loop control systems (artificial pancreas) behaving as if the control gain is increased and the target is lowered. In this arm we study closed-loop control with a sensor signal reading equal to blood glucose.
- LOW Error: Glucose sensor errors leading to sensor glucose reading higher than that true blood glucose result in closed-loop control systems (artificial pancreas) behaving as if the control gain is increased and the target is lowered. In this arm we study closed-loop control with a sensor signal reading 20% lower than blood glucose.
Arm/Group | HIGH Error | NO Error | LOW Error
Number analyzed (Participants) | 5 | 5 | 5
mmol/l/min | 66.8 [53.3 to 80.3] | 48.8 [41.1 to 56.4] | 37.4 [33.4 to 41.5]
Statistical Analysis 1: Comparison: HIGH Error vs NO Error vs LOW Error; Differences among the 3 groups were assessed by repeated measures ANOVA using Sidak's correction for multiple comparisons. All subjects were analyzed as a single group, no comparison group; Test type: Other — ANOVA was used to first tests the hypothesis that there is a difference among the three groups; p = 0.0011, ANOVA — The p value was adjusted for multiple comparisons using Sidak's correction. A priori the pimary outcome was defined as blood glucose AUC from 8 am - 12pm; however we used blood glucose AUC from 8am - 2pm to capture the entire meal response; Mean Difference (Final Values) = 66.8, 95% CI 2-sided [33.4 to 80.3]

2. Secondary Outcome: Peak and Nadir Postprandial Glucose Concentration
Description: Highest and lowest glucose concentrations obtained during breakfast meal.
Time Frame: On day #1, day #2 and day #3 (each day could be 24 hours to 7 days apart from prior one, and completed within 6 week period) 8:00 AM to 12:00 PM on day following admission, with samples obtained every 10-15 minutes, for each sequence of calibration errors
Population: Analysis was limited to the 5 subjects completed all aspects of the study per protocol (i.e. 5 subjects who completed all three scheduled breakfast meals).
Measure: Mean (95% Confidence Interval); unit: mmol/l
Groups:
- Gain Increased and Target Decreased; Nadir Mean: Closed-loop control performed with a sensor reading higher than blood glucose behave as if the control gain has been increased and the target set lowered
- Gain Decreased and Target Increased: Closed-loop control performed with a sensor reading lower than blood glucose behave as if the control gain has been lowered and the target increased
Arm/Group | Gain Increased and Target Decreased | Nadir Mean | Gain Decreased and Target Increased
Number analyzed (Participants) | 5 | 5 | 5
mmol/l
  Peak glucose concentration | 13.3 [11.3 to 15.4] | 11.8 [9.8 to 14.0] | 11.3 [10.2 to 12.4]
  Nadir glucose concentration | 4.5 [3.8 to 5.2] | 4.8 [3.7 to 6.5] | 6.6 [5.6 to 7.5]
Statistical Analysis 1: Comparison: Gain Increased and Target Decreased; Test type: Other; p = 0.0059, ANOVA

3. Other Pre Specified Outcome: Nighttime Time-in-target 5.0-8.33mmol/l (Controller Set-point Plus and Minus 15 mg/dL)
Description: Night-time in target range 5.0-8.33, following the 3 hour controller initialization period blood glucose remained at or near target.
Time Frame: On day #1, day #2 and day #3 (each day could be 24 hours to 7 days apart from prior one, and completed within 6 week period) 12:00 AM to 6:00 AM on day following admission, with samples obtained every 10-15 minutes, for each sequence of calibration errors
Population: Analysis was limited to the 6 subjects completing all 3 nighttime periods per protocol
Measure: Median (Inter-Quartile Range); unit: percentage of time in target range
Groups:
- HIGH Error: Closed-loop control performed with sensor glucose reading higher than blood glucose behaves as if the controller gain has been increased and the target lowered
- NO Errror: Reference nighttime response for comparison with closed-loop control with sensor glucose reading higher than blood glucose and lower than blood glucose.
- LOW Error: Closed-loop control performed with sensor glucose reading lower than blood glucose behaves as if the controller gain has been lowered and the target increased
Arm/Group | HIGH Error | NO Errror | LOW Error
Number analyzed (Participants) | 6 | 6 | 6
percentage of time in target range | 88 [87 to 100] | 100 [100 to 100] | 80 [54 to 86]

ADVERSE EVENTS:
Time Frame: Study data was collected over a 6 month period, in the Center for Clinical Investigations at the Beth Israel Deaconess Medical Center
Description: Adverse events were to be reported to the CCI in accordance with CCI policy (Section XII, G of the CCI Policy and Procedure manual) on reporting such events
Groups:
- HIGH Error First, NO Error Second, LOW Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control calculated to be 33% higher than the true glucose (HIGH error), then with the value equal to the true glucose (NO error), and then with the value calculated to be 80% of the true value (LOW error).
- HIGH Error First, LOW Error Second, NO Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control calculated to be 33% higher than the true glucose (HIGH error), then with the value calculated to be 80% of the true value (LOW error), and then with the value equal to the true glucose (NO error).
- NO Error First, HIGH Error Second, LOW Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control equal to the true glucose (NO error), then with the value calculated to be 33% higher than the true glucose (HIGH error), and then with the value calculated to be 80% of the true value (LOW error).
- NO Error First, LOW Error Second, HIGH Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control equal to the true glucose (NO error), then with the value calculated to be 80% of the true value (LOW error) and then with the value calculated to be 33% higher than the true glucose (HIGH error)
- LOW Error First, NO Error Second, HIGH Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control equal 80% of the true value (LOW error), then with value equal to the true glucose (NO error), and then with the value calculated to be calculated to be 33% higher than the true glucose (HIGH error).
- LOW Error First, HIGH Error Second, NO Error Third: Nighttime and Breakfast closed-loop glucose control was performed on 3 occasions: first with the glucose value used for control calculated to be 20% lower than the true glucose (LOW error), then with the value calculated to be 30% higher than the true value (HIGH error) and then with the value equal to the true glucose (NO error)
Arm/Group | HIGH Error First, NO Error Second, LOW Error Third | HIGH Error First, LOW Error Second, NO Error Third | NO Error First, HIGH Error Second, LOW Error Third | NO Error First, LOW Error Second, HIGH Error Third | LOW Error First, NO Error Second, HIGH Error Third | LOW Error First, HIGH Error Second, NO Error Third
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
In this study sensor calibration errors were simulated using a YSI reference glucose values; however, this may not fully capture errors that are due to delays between plasma and the interstitial fluid glucose value measured by a glucose sensor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No